CLINICAL TRIAL: NCT02449317
Title: Bioimpedance Analysis Guided Volume Expansion for the Prevention of Contrast
Brief Title: Bioimpedance Analysis Guided Volume Expansion for the Prevention of Contrast Induced-acute Kidney Injury
Acronym: BELIEVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2558/171
Record Dates: First submitted 2015-05-17; First posted 2015-05-20 (Estimated); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: X-ray Contrast Media Adverse Reaction
Keywords: contrast induced acute kidney injury; bioimpedance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Other): standard hydration : 7.5% Sodium bicarbonate 150 ml + 5% dextrose in water 850 ml IV 1 ml/kg/hr in 6 hours
  Interventions: Other: standard hydration
- Bioimpedance guided (Experimental): Bioelectrical impedance analysis guided hydration therapy : 7.5% Sodium bicarbonate 150 ml + 5% dextrose in water 850 ml IV in 6 hours rate was adjusted regarding to extracellular water/total body water
  * extracellular water/total body water < 0.36 : 4 ml/kg/hr
  * extracellular water/total body water 0.36-0.4 : 2 ml/kg/hr
  * extracellular water/total body water > 0.4 : 1 ml/kg/hr
  Interventions: Other: Bioimpedance guided

INTERVENTIONS:
Other: Bioimpedance guided — bioelectrical impedance analysis guided hydration therapy : 7.5% Sodium bicarbonate 150 ml + 5% dextrose in water 850 ml IV in 6 hours rate was adjusted regarding to extracellular water/total body water
  * extracellular water/total body water < 0.36 : 4 ml/kg/hr
  * extracellular water/total body water 0.36-0.4 : 2 ml/kg/hr
  * extracellular water/total body water > 0.4 : 1 ml/kg/hr
  Arms: Bioimpedance guided
Other: standard hydration — standard hydration : 7.5%Sodium bicarbonate 150 ml + 5% dextrose in water 850 ml IV 1 ml/kg/hr in 6 hours
  Arms: Control

SUMMARY:
Bioelectrical impedance analysis guided volume expansion for the prevention of contrast induced-acute kidney injury

DETAILED DESCRIPTION:
Compared bioelectrical impedance analysis guided hydration therapy versus standard hydration for the prevention of contrast induced-acute kidney injury

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-90 yr
2. Chronic kidney disease stage 3 & 4 (eGFR 15-60 ml/min/m2)
3. elective cardiac catheterization

Exclusion Criteria:

1. Contrast media administration in the past 14 days
2. congestive heart failure (NYHA III-IV, ascites , pleuropericardial effusion ,severe valvular heart disease
3. Kidney transplant status or RRT
4. Emergency cardiac catheterization
5. Allergy to radiographic contrast media
6. Unstable renal function (change in serum creatinine ≥ 0.5 mg/dl or 25% within 14 days prior to the study
7. Not inform consent
8. left ventricular ejection fraction < 40 %
9. Liver cirrhosis child B or C
10. Dosage of angiotensin-converting enzyme inhibitor /angiotensin II receptor blocker changed in past 2 wk

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
serum creatinine at 48-72 hours after contrast administration | 48-72 hr
  Acute kidney injury

SECONDARY OUTCOMES:
serum creatinine at 2 weeks after contrast administration | 2 weeks
  Renal replacement therapy

CONTACTS AND LOCATIONS:
Overall Officials: Arkom Nongnuch, MD, Principal Investigator — Ramathibodi hospital, Mahidol university